CLINICAL TRIAL: NCT02251301
Title: The Effect of Adding Milk in Proximity to Exercise During an Interval Training Intervention in Type 2 Diabetes (T2D) on Metabolic and Cardiovascular Health.
Brief Title: Milk Plus Exercise: A Novel Strategy to Treat Diabetes.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Dairy Farmers of Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: H14-01636
Record Dates: First submitted 2014-09-25; First posted 2014-09-29 (Estimated); Last update posted 2017-05-02 (Actual); Status verified 2016-08

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — High-Intensity Interval Training; Water; Proteins

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Macronutrient isoenergetic control (Active Comparator): Participants will also engage in twelve weeks of high intensity interval training with consumption of one serving (250 mL) of macro nutrient matched isoenergetic control (whey/casein protein and dextrose/lactose) consumed immediately and 1 h after each training session
  Interventions: Behavioral: High intensity interval training; Dietary Supplement: Macronutrient isoenergetic control
- Skim Milk (Experimental): Participants will also engage in twelve weeks of High intensity interval training with consumption of one serving (250 mL) of fat-free fluid milk immediately and 1 h after each training session
  Interventions: Dietary Supplement: Skim Milk; Behavioral: High intensity interval training
- Placebo (Placebo Comparator): Participants will also engage in twelve weeks of high intensity interval training with consumption of one serving (250 mL) of placebo (water) consumed immediately and 1 h after each training session.
  Interventions: Behavioral: High intensity interval training; Other: Placebo

INTERVENTIONS:
Dietary Supplement: Skim Milk — 250 ml skim milk will be consumed by participants immediately and 1 hour after each of the 36 sessions of high-intensity interval training over a 12 week period.
  Other Names: Fat-free milk
  Arms: Skim Milk
Behavioral: High intensity interval training — All participants will undergo a 12 week high intensity interval training program consisting of 3 supervised sessions a week of 4-10 x 1 min high intensity interval alternating with 1 min of recovery.
Other: Placebo — 250 mL water will be consumed by participants immediately and 1 hour after each of the 36 sessions of high-intensity interval training over a 12 week period.
  Other Names: water
  Arms: Placebo
Dietary Supplement: Macronutrient isoenergetic control — 250 mL of protein+cho matched drink will be consumed by participants immediately and 1 hour after each of the 36 sessions of high-intensity interval training over a 12 week period.
  Other Names: Protein
  Arms: Macronutrient isoenergetic control

SUMMARY:
The purpose of this study is to investigate whether combining interval training with skim milk supplementation will result in improved glucose control and markers of cardiovascular health in people with type 2 diabetes. Participants will complete supervised interval training three times a week over a 12 week training period while consuming skim-milk, whey/casein protein drink, or a placebo beverage that does not contain any calories or vitamins/minerals immediately and 1 hour after each training session. After twelve weeks participants will repeat baseline tests to examine any effects of the intervention on their glucose control, fitness, blood vessel function, body composition, and blood markers of inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 40 and 75.
* Diagnosed with type 2 diabetes for more than 6 months.
* On stable medication for the last 6 months

Exclusion Criteria:

* Type 2 diabetes controlled with exogenous insulin
* Uncontrolled hypertension (blood pressure >160/90 mmHg)
* History of heart disease, myocardial infarction or stroke
* Any other contraindications to exercise

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2015-01; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in glycemic control assessed by continuous glucose monitoring at end of week 12 of intervention | Baseline, Week 12.

SECONDARY OUTCOMES:
Change from baseline in hemoglobin A1C percentage at end of week 12 of intervention. | Baseline, Week 12.
Change from baseline in fasting plasma glucose concentration at end of week 12 of intervention. | Baseline, Week 12.
Change from baseline in fasting plasma insulin concentration at end of week 12 of intervention. | Baseline, Week 12.
Change from baseline in flow mediated dilation of brachial artery at end of week 12 of intervention. | Baseline, Week 12.
Change from baseline in peak oxygen uptake as a measure of aerobic fitness at end of week 12 of intervention. | Baseline, Week 12

OTHER OUTCOMES:
Change from baseline in fasting plasma non esterified free fatty acid concentration at end of week 12 of intervention. | Baseline, Week 12
Change from baseline in systolic blood pressure at end of week 12 of intervention. | Baseline, Week 12
Change from baseline in diastolic blood pressure at end of week 12 of intervention. | Baseline, Week 12.
Change from baseline in circulating inflammatory cytokines at end of week 12 of intervention. | Baseline, Week 12.
Change from baseline in body composition as measured by dual absorbancy x ray at end of week 12 of intervention. | Baseline, Week 12.
Change from baseline in task switching capabilities at end of week 12 of intervention. | Baseline, Week 12.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan P Little, PHD, Principal Investigator — University of British Columbia
Locations (1):
- University of British Columbia, Okanagan., Kelowna, British Columbia, Canada

REFERENCES:
- [Derived] Francois ME, Pistawka KJ, Halperin FA, Little JP. Cardiovascular benefits of combined interval training and post-exercise nutrition in type 2 diabetes. J Diabetes Complications. 2018 Feb;32(2):226-233. doi: 10.1016/j.jdiacomp.2017.10.002. Epub 2017 Nov 29. PMID 29198993